CLINICAL TRIAL: NCT04419701
Title: Comparison of Ultrasound Guided Genicular Nerve Block and Periarticular Infiltration for Postoperative Pain in Knee Arthroplasty
Brief Title: Comparison of Ultrasound Guided Genicular Nerve Block and Periarticular Infiltration in Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: pain in knee arthroplasty
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- periarticular infiltration group (Experimental): will receive intraoperative periarticular infitration consisting of 89.5 mL of normal saline, 20 mL of 5% bupivacaine and 0.5 mL of adrenaline (4.5 ugm/ml) with a concentration 1:220000 (total volume: 110 mL)
  Interventions: Procedure: periarticular infiltration
- genicular nerve block group (Experimental): will receive ultrasound guided genicular nerve block at three nerves, i.e., superomedial, superolateral, and inferomedial genicular nerves consisting of 15 ml bupivacaine 0.25% with adrenaline 2.5 µg/ml with a concentration 1:400000 in the immediate postoperative period.
  Interventions: Procedure: genicular nerve block

INTERVENTIONS:
Procedure: periarticular infiltration — The cocktail will be injected at the following 7 anatomical zones as follows:
  Zone 1: medial retinaculum Zone 2: medial collateral ligament and medial meniscus capsular attachment Zone 3: posterior capsule Zone 4: lateral collateral ligament and lateral meniscus capsular attachment Zone 5: lateral retinaculum Zone 6: patellar tendon and fat pad Zone 7: cut ends of quadriceps muscle and tendon Injection at zones 2, 3, and 4 will be administered after making the tibial and femoral cuts and ligament balancing. At zones 1, 5, 6, and 7, the injection will be administered after implant placement.
  Arms: periarticular infiltration group
Procedure: genicular nerve block — The genicular arteries will be identified near the periosteal areas, which are the junctions of the epicondyle and the shafts of the femur and tibia, and confirmed by color Doppler ultrasound. genicular nerve block target points should be next to each genicular artery because the superior lateral, superior medial, and inferior medial genicular artery traveled along each genicular nerve.After using color Doppler to confirm the genicular artery, the needle will be inserted in the plane of the ultrasound probe in the long-axis view.
  Arms: genicular nerve block group

SUMMARY:
Effective pain relief allows the patients to obtain early knee mobilization and optimal rehabilitation and thus improves the patient satisfaction.

The aim of perioperative pain control is to minimize delays in recovery, postoperative delirium and pain-related stress responses that can lead to serious morbidity and poor outcomes. Numerous approaches to effectively control postoperative pain in TKA patients have been evaluated, as poorly controlled acute postoperative pain can be associated with persistent pain. Furthermore, increased pain intensity after surgery on the second knee seems to be closely associated with chronic post-TKA pain, with similar mechanisms underlying hyperalgesia or chronic pain.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA), one of the most commonly performed operations in orthopaedic department, has been a successful intervention for patients with end-stage knee arthritis.

Rehabilitation after total knee arthroplasty (TKA) routinely starts immediately after surgery on the postoperative ward and therefore requires adequate analgesia. An ideal analgesic modality for post-TKA rehabilitation should permit adequate knee flexion with minimal pain without motor impairment, resulting in successful mobilization. Pain control plays an essential role in the overall postoperative period for the patients undergoing TKA.

Effective pain relief allows the patients to obtain early knee mobilization and optimal rehabilitation and thus improves the patient satisfaction.

The aim of perioperative pain control is to minimize delays in recovery, postoperative delirium and pain-related stress responses that can lead to serious morbidity and poor outcomes. Numerous approaches to effectively control postoperative pain in TKA patients have been evaluated, as poorly controlled acute postoperative pain can be associated with persistent pain. Furthermore, increased pain intensity after surgery on the second knee seems to be closely associated with chronic post-TKA pain, with similar mechanisms underlying hyperalgesia or chronic pain.

Traditionally, the degree of knee flexion has been used as an outcome measure after TKA to evaluate functional recovery and the success of the type of analgesia used.

Several methods such as intravenous opioids, extraarticular and intraarticular injection, epidural analgesia and femoral or sciatic nerve blocks are currently used for postoperative pain management.

However, each method is reported with potential side effects, for example, opioid drugs caused vomiting, nausea, constipation, dizziness and urinary retention, epidural analgesia with urinary retention, respiratory depression and spinal headache, femoral or sciatic block with diminished muscle control and possible nerve damage.

Periarticular multimodal drug injection in TKA is a technique that patients received intraoperative drug injection in the periarticular fields such as posterior capsule, medial and lateral collateral ligaments, quadriceps mechanism and peripatellar tissue at the end of the surgery. Multimodal drugs mainly consist of local anaesthetics, non-steroidal anti-inflammatory drugs, opioids, epinephrine with or without corticosteroid.

Genicular nerve block (GNB) and ablation have been used for managing chronic pain from knee osteoarthritis with good success.

ELIGIBILITY:
Inclusion Criteria:

* unilateral knee arthroplasty surgery,
* aged more than 50 years of both genders.
* have american society of anesthesiologist physical status I-II and III.

Exclusion Criteria:

* Revision knee arthroplasty,
* previous surgery or trauma to knee,
* drug allergy, regular narcotic use,
* renal impairments
* hepatic impairments,
* neuromuscular diseases
* coagulopathy disorders.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
total doses of postoperative opioid consumption | postoperative first day
  total doses of postoperative rescue morphine consumption

SECONDARY OUTCOMES:
Time of the first dose of rescue analgesia | postoperative first day
  Time of the first dose of rescue morphine analgesia at dose of 3 mg

OTHER OUTCOMES:
Knee range of motion | postoperative first day
  The knee primarily only moves in one plane of movement, flexion and extension. A completely straight knee joint will measure 0° and a fully bent knee will have a flexion of at 135° degrees
Knee range of motion | postoperative second day
  The knee primarily only moves in one plane of movement, flexion and extension. A completely straight knee joint will measure 0° and a fully bent knee will have a flexion of at 135° degrees
Knee range of motion | postoperative third day
  The knee primarily only moves in one plane of movement, flexion and extension. A completely straight knee joint will measure 0° and a fully bent knee will have a flexion of at 135° degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek Abdel Hay, Tanta, El Gharbyia, Egypt